CLINICAL TRIAL: NCT02334982
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Safety, Tolerability and Pharmacokinetic Study of Escalating Single Doses of TAK-137 in Healthy Subjects
Brief Title: Safety, Tolerability and Pharmacokinetics of Escalating Single Doses of TAK-137 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: TAK-137_101; U1111-1164-7376 (Registry Identifier: WHO)
Record Dates: First submitted 2015-01-06; First posted 2015-01-09 (Estimated); Results first posted 2015-02-10 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-01

CONDITIONS: Dose Finding Study
Keywords: Drug therapy
MeSH Terms: interventions — TAK-137

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Cohort 1: TAK-137 2 mg (Experimental): TAK-137 2 mg, tablets, orally, once on Day 1.
  Interventions: Drug: TAK-137
- Cohort 2: TAK-137 5 mg (Experimental): TAK-137 5 mg, tablets, orally, once on Day 1.
  Interventions: Drug: TAK-137
- Cohort 3: TAK-137 10 mg (Experimental): TAK-137 10 mg, tablets, orally, once on Day 1.
  Interventions: Drug: TAK-137
- Cohort 4: TAK-137 5 mg Food Effect (Experimental): TAK-137 5 mg, tablets, orally, under fasted conditions, once on Day 1 of Period 1, followed by 14 days of follow-up, followed by TAK-137 5 mg, tablets, orally, under fed conditions, once on Day 1 of Period 2.
  Interventions: Drug: TAK-137
- Cohort 5: TAK-137 0.5 mg (Experimental): TAK-137 0.5 mg, tablets, orally, once on Day 1.
  Interventions: Drug: TAK-137
- Cohort 6: TAK-137 20 mg (Experimental): TAK-137 20 mg, tablets, orally, once on Day 1.
  Interventions: Drug: TAK-137
- Cohorts 1-6: Placebo (Placebo Comparator): TAK-137 placebo-matching tablets, orally, once on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAK-137 — TAK-137 tablets
  Arms: Cohort 1: TAK-137 2 mg; Cohort 2: TAK-137 5 mg; Cohort 3: TAK-137 10 mg; Cohort 4: TAK-137 5 mg Food Effect; Cohort 5: TAK-137 0.5 mg; Cohort 6: TAK-137 20 mg
Drug: Placebo — TAK-137 placebo-matching tablets
  Arms: Cohorts 1-6: Placebo

SUMMARY:
The purpose of this study is to characterize the safety and tolerability profile of TAK-137 when administered as a single dose of tablets at escalating dose levels in healthy participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-137. TAK-137 is being tested to find a safe and well-tolerated dose. This study looked at safety (lab results and side effects) and pharmacokinetic properties (drug absorption, distribution, metabolism, and excretion) in people who took TAK-137. This study was designed as a single ascending 6 Cohort dose study with planned doses of 2, 5, 15, 50, and 100 mg and Cohort 6 dose to be determined if the maximum tolerated dose (MTD) was not reached. Anticipated enrollment was 48.

This study enrolled 47 participants and consisted of 6 Cohorts. Participants in Cohorts 1, 2, 3, 5 and 6 were randomized to receive a single dose of TAK-137 or placebo after a 10-hour fast. Participants in Cohort 4 were randomized to receive a single dose of TAK-137 or placebo under fasted conditions, followed by a single dose of TAK-137 or placebo under fed conditions 14 days later. Participants in cohort 4 will receive the same dose in both fasted and fed conditions. The starting dose was 2 mg followed by administrations of 5, 10, 0.5 and 20 mg.

This single-center trial was conducted in the United States. For Cohorts 1, 2, 3, 5, and 6 the overall time to participate in this study was up to 42 days. Participants made 4 visits to the clinic including one 5-day period of confinement to the clinic, and were contacted by telephone 14 days after last dose of study drug for a follow-up assessment.

For Cohort 4 the overall time to participate in this study was up to 56 days. Participants made 7 visits to the clinic including two 5-day periods of confinement to the clinic, and were contacted by telephone 14 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy male or non-pregnant, non-lactating female adult who is 18 to 55 years of age inclusive at the time of informed consent and first study medication dose.
2. Weighs at least 45 kg and has a body mass index (BMI) between 18 and 30.0 kg/m^2, inclusive at Screening.
3. Is able to comply with the protocol and is willing to sign the informed consent prior to undergoing any study-related procedures.

Exclusion Criteria:

1. Has a known hypersensitivity to any component of the formulation of TAK-137.
2. Has a medical condition such as mental retardation that can cause cognitive impairment.
3. Has a risk of suicide according to the Investigator's clinical judgment (eg, per Columbia-Suicide Severity Rating Scale [C-SSRS] or has made a suicide attempt in the previous 6 months).
4. Has evidence of current cardiovascular, central nervous system, hepatic, hematopoietic disease, renal dysfunction, metabolic or endocrine dysfunction, serious allergy, asthma hypoxemia, hypertension, seizures, or allergic skin rash.
5. There is any finding in the participant's medical history, physical examination, or safety laboratory tests (including safety electroencephalogram [EEG]) giving reasonable suspicion of a disease that would contraindicate taking TAK-137, or a similar drug in the same class, or that might interfere with the conduct of the study. This includes, but is not limited to, peptic ulcer disease, seizure disorders, and cardiac arrhythmias.
6. Has taken any excluded medication, supplements, or food products listed in the Excluded Medications and Dietary Products table.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2013-06; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 21 June 2013 to 30 January 2014.
Pre-assignment Details: Healthy Volunteers were enrolled in a 6 Cohort randomized, dose escalating study at doses of 0.5, 2,5, 10 and 20 mg TAK-137 tablets or placebo single dose once in Cohorts 5,1,2,3 and 6 fasting respectively. Cohort 4 received 5 mg tablets or placebo single dose fasting then 5 mg or placebo fed.
Period: Overall Study
Arm/Group | Cohort 1: TAK-137 2 mg | Cohort 2: TAK-137 5 mg | Cohort 3: TAK-137 10 mg | Cohort 4: TAK-137 5 mg Food Effect | Cohort 5: TAK-137 0.5 mg | Cohort 6: TAK-137 20 mg | Cohorts 1-6: Placebo
Started | 6 | 5 | 6 | 6 | 6 | 6 | 12
Completed | 6 | 5 | 6 | 6 | 6 | 6 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: TAK-137 2 mg | Cohort 2: TAK-137 5 mg | Cohort 3: TAK-137 10 mg | Cohort 4: TAK-137 5 mg Food Effect | Cohort 5: TAK-137 0.5 mg | Cohort 6: TAK-137 20 mg | Cohorts 1-6: Placebo | Total
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 12 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (9.00) | 34.0 (8.66) | 40.5 (8.22) | 36.5 (9.27) | 24.7 (3.88) | 38.5 (10.63) | 31.5 (6.87) | 34.9 (9.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 2 | 4 | 5 | 6 | 20
  Male | 4 | 4 | 6 | 4 | 2 | 1 | 6 | 27
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 4
  Black or African American | 1 | 3 | 2 | 2 | 3 | 3 | 5 | 19
  White | 4 | 1 | 3 | 4 | 2 | 3 | 5 | 22
  Multiracial | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 3 | 1 | 3 | 1 | 3 | 1 | 3 | 15
  Non-Hispanic or Latino | 3 | 4 | 3 | 5 | 3 | 5 | 9 | 32
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 6 | 6 | 6 | 6 | 12 | 47
Height [Mean (Standard Deviation); unit: cm] | 170.3 (8.19) | 173.2 (13.22) | 178.0 (6.63) | 172.3 (8.62) | 171.5 (6.44) | 164.7 (11.74) | 166.2 (9.44) | 171.6 (9.52)
Weight [Mean (Standard Deviation); unit: kg] | 70.97 (15.299) | 79.86 (14.870) | 81.88 (15.381) | 74.40 (18.840) | 75.05 (12.228) | 64.18 (14.297) | 73.23 (9.378) | 74.23 (15.306)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.22 (3.276) | 26.48 (2.138) | 25.68 (3.323) | 24.68 (4.260) | 25.38 (2.905) | 23.38 (2.315) | 26.51 (2.658) | 24.93 (3.074)
Caffeine Consumption [Number; unit: participants]
  Yes | 0 | 1 | 2 | 2 | 1 | 1 | 5 | 12
  No | 6 | 4 | 4 | 4 | 5 | 5 | 7 | 35
Smoking Classification [Number; unit: participants]
  Never smoked | 6 | 5 | 6 | 5 | 6 | 6 | 12 | 46
  Ex-smoker | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Alcohol Classification [Number; unit: participants]
  Never | 6 | 5 | 4 | 5 | 6 | 6 | 12 | 44
  Current | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced at Least 1 Treatment-Emergent Adverse Event
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Day 1 to 14 days after the last dose of study medication(Up to 30 days)
Population: Safety population included all participants who received at least one dose of study medication. 8 of the 47 enrolled participants participated in Cohort 4 fed.
Measure: Number; unit: percentage of participants
Groups:
- TAK-137 0.5 mg: TAK-137 0.5 mg, tablets, orally, fasting, once on Day 1.
- TAK-137 2 mg: TAK-137 2 mg, tablets, orally, fasting, once on Day 1.
- TAK-137 5 mg (Fasting): TAK-137 5 mg, tablets, orally, fasting, once on Day 1.
- TAK-137 10 mg: TAK-137 10 mg, tablets, orally, once on Day 1.
- TAK-137 20 mg: TAK-137 20 mg, tablets, orally, fasting, once on Day 1.
- TAK-137 Placebo: TAK-137 placebo-matching tablets, orally, once on Day 1.
- TAK-137 5 mg (Fed): TAK-137 5 mg, tablets, orally, fed, once, on Day 1 of Period 2.
- Placebo (Fed): TAK-137 placebo-matching tablets, orally, fed, once on Day 1of Period 2.
Arm/Group | TAK-137 0.5 mg | TAK-137 2 mg | TAK-137 5 mg (Fasting) | TAK-137 10 mg | TAK-137 20 mg | TAK-137 Placebo | TAK-137 5 mg (Fed) | Placebo (Fed)
Number analyzed (Participants) | 6 | 6 | 11 | 6 | 6 | 12 | 6 | 2
percentage of participants | 0 | 16.7 | 0 | 16.7 | 50.0 | 33.3 | 16.7 | 0

2. Primary Outcome: Percentage of Participants With Abnormal Safety Laboratory Findings
Description: The percentage of participants with any markedly abnormal standard safety laboratory values was collected throughout study.
Time Frame: Day 1 to 14 days after the last dose of study medication (Up to 30 Days)
Population: Participants from the Safety population, all participants who received at least one dose of study medication, with data available for analysis. 8 of the 47 enrolled participants participated in Cohort 4 fed.
Measure: Number; unit: percentage of participants
Groups:
- Placebo Fasting: TAK-137 placebo-matching tablets, orally, fasting, once on Day 1.
Arm/Group | TAK-137 0.5 mg | TAK-137 2 mg | TAK-137 5 mg (Fasting) | TAK-137 10 mg | TAK-137 20 mg | Placebo Fasting | TAK-137 5 mg (Fed) | Placebo (Fed)
Number analyzed (Participants) | 6 | 6 | 11 | 6 | 6 | 12 | 6 | 2
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Percentage of Participants With Markedly Abnormal Vital Sign Measurements
Description: The percentage of participants with any markedly abnormal standard vital sign measurements was collected throughout study.
Time Frame: Day 1 to 14 days after the last dose of study medication
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Groups:
- TAK-137 Placebo: TAK-137 placebo-matching tablets, orally, fasting, once on Day 1.
Arm/Group | TAK-137 0.5 mg | TAK-137 2 mg | TAK-137 5 mg (Fasting) | TAK-137 10 mg | TAK-137 20 mg | TAK-137 Placebo | TAK-137 5 mg (Fed) | Placebo (Fed)
Number analyzed (Participants) | 6 | 6 | 11 | 6 | 6 | 12 | 6 | 2
percentage of participants
  Pulse (5 min after supine) <50 bpm | 0 | 16.7 | 0 | 16.7 | 0 | 8.3 | 0 | 0
  Pulse (5 min after supine) >120 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse (1 min after standing) <50 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse (1 min after standing) >120 bpm | 0 | 0 | 0 | 16.7 | 0 | 8.3 | 16.7 | 0
  Pulse (3 min after standing) <50 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse (3 min after standing) >120 bpm | 0 | 0 | 0 | 0 | 0 | 8.3 | 16.7 | 0
  Systolic BP (5 min after supine) <85 mmHG | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0
  Systolic BP (5 min after supine) >180 mmHG | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Systolic BP (1 min after standing) <85 mmHG | 0 | 16.7 | 0 | 0 | 50.0 | 0 | 0 | 0
  Systolic BP (1 min after standing) >180 mmHG | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Systolic BP (3 min after standing) <85 mmHG | 0 | 16.7 | 9.1 | 0 | 16.7 | 0 | 0 | 0
  Systolic BP (3 min after standing) >180 mmHG | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Diastolic BP (5 min after supine) <50 mmHg | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0
  Diastolic BP (5 min after supine) >110 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Diastolic BP (1 min after standing) <50 mmHg | 0 | 16.7 | 0 | 0 | 16.7 | 0 | 0 | 0
  Diastolic BP (1 min after standing) >110 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Diastolic BP (3 min after standing) <50 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Diastolic BP (3 min after standing) >110 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-137
Description: Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Time Frame: Day 1
Population: Participants from the Pharmacokinetic (PK) set, all participants who receive study drug and have at least one measureable concentration, with data available for analysis of this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Cohort 1: TAK-137 2 mg: TAK-137 2 mg, tablets, orally, fasting, once on Day 1.
- Cohort 2: TAK-137 5 mg (Fasting): TAK-137 5 mg, tablets, orally, fasting, once on Day 1.
- Cohort 4: TAK-137 5 mg (Fasting): TAK-137 5 mg, tablets, orally, fasting, once on Day 1 of Period 1.
- Cohort 5: TAK-137 0.5 mg: TAK-137 0.5 mg, tablets, orally, fasting, once on Day 1.
- Cohort 6: TAK-137 20 mg: TAK-137 20 mg, tablets, orally, fasting, once on Day 1.
- Cohort 4: TAK-137 5 mg (Fed): TAK-137 5 mg, tablets, orally, fed, once, on Day 1 of Period 2.
Arm/Group | Cohort 1: TAK-137 2 mg | Cohort 2: TAK-137 5 mg (Fasting) | Cohort 3: TAK-137 10 mg | Cohort 4: TAK-137 5 mg (Fasting) | Cohort 5: TAK-137 0.5 mg | Cohort 6: TAK-137 20 mg | Cohort 4: TAK-137 5 mg (Fed)
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 6
ng/mL | 38.8 (8.64) | 68.90 (7.40) | 121.1 (28.44) | 61.1 (16.11) | 9.0 (0.76) | 206.1 (80.72) | 85.9 (28.58)

5. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-137
Description: Time to reach the maximum plasma concentration (Cmax), equal to time (hours) to Cmax.
Time Frame: Day 1
Population: as for outcome 4
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: TAK-137 2 mg | Cohort 2: TAK-137 5 mg (Fasting) | Cohort 3: TAK-137 10 mg | Cohort 4: TAK-137 5 mg (Fasting) | Cohort 5: TAK-137 0.5 mg | Cohort 6: TAK-137 20 mg | Cohort 4: TAK-137 5 mg (Fed)
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 6
hours | 2.00 [1.00 to 3.00] | 3.00 [1.50 to 6.00] | 3.00 [2.00 to 8.00] | 2.50 [1.00 to 3.00] | 2.00 [1.00 to 3.00] | 2.50 [1.50 to 6.00] | 5.50 [2.00 to 12.00]

6. Secondary Outcome: AUC(0-tlqc): Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-137
Description: (AUC(0-tlqc) is a measure of total plasma exposure to the drug from Time 0 to Time of the Last Quantifiable Concentration (AUC[0-tlqc]).
Time Frame: Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Cohort 1: TAK-137 2 mg | Cohort 2: TAK-137 5 mg (Fasting) | Cohort 3: TAK-137 10 mg | Cohort 4: TAK-137 5 mg (Fasting) | Cohort 5: TAK-137 0.5 mg | Cohort 6: TAK-137 20 mg | Cohort 4: TAK-137 5 mg (Fed)
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 6
ng*hr/mL | 405 (121.6) | 1668 (787.6) | 3012 (2204.1) | 1191 (767.9) | 94 (41.9) | 5346 (3292.4) | 1470 (434.5)

7. Secondary Outcome: AUC(0-inf): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-137
Description: AUC(0-inf) is a measure of total plasma exposure to the drug from time zero extrapolated to infinity.
Time Frame: Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Cohort 1: TAK-137 2 mg | Cohort 2: TAK-137 5 mg (Fasting) | Cohort 3: TAK-137 10 mg | Cohort 4: TAK-137 5 mg (Fasting) | Cohort 5: TAK-137 0.5 mg | Cohort 6: TAK-137 20 mg | Cohort 4: TAK-137 5 mg (Fed)
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 6
ng*hr/mL | 408 (121.64) | 1696 (803.9) | 3135 (2380.8) | 1198 (766.64) | 97 (43.24) | 5353 (3295.2) | 1474 (436.1)

8. Secondary Outcome: Terminal Elimination Half-life (T1/2) for TAK-137_101
Description: Terminal Phase Elimination Half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma.
Time Frame: Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1: TAK-137 2 mg | Cohort 2: TAK-137 5 mg (Fasting) | Cohort 3: TAK-137 10 mg | Cohort 4: TAK-137 5 mg (Fasting) | Cohort 5: TAK-137 0.5 mg | Cohort 6: TAK-137 20 mg | Cohort 4: TAK-137 5 mg (Fed)
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 6
hours | 6.65 (2.462) | 12.66 (2.491) | 13.60 (7.105) | 15.77 (10.553) | 8.54 (4.487) | 13.09 (5.276) | 10.52 (3.875)

9. Secondary Outcome: Apparent Clearance (CL/F) for TAK-137_101
Description: CL/F is apparent clearance of the drug from the plasma, calculated as the drug dose divided AUC(0-inf), expressed in liters per hour (L/hr).
Time Frame: Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: liters/hour
Arm/Group | Cohort 1: TAK-137 2 mg | Cohort 2: TAK-137 5 mg (Fasting) | Cohort 3: TAK-137 10 mg | Cohort 4: TAK-137 5 mg (Fasting) | Cohort 5: TAK-137 0.5 mg | Cohort 6: TAK-137 20 mg | Cohort 4: TAK-137 5 mg (Fed)
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 6
liters/hour | 5.22 (1.304) | 3.66 (1.912) | 5.23 (3.877) | 5.91 (3.372) | 6.26 (3.062) | 7.19 (6.976) | 3.63 (0.996)

10. Secondary Outcome: Apparent Volume of Distribution (Vz/F) for TAK-137_101
Description: Vz/F is the distribution of a drug between plasma and the rest of the body following oral administration, calculated as CL/F divided by λz.
Time Frame: Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Cohort 1: TAK-137 2 mg | Cohort 2: TAK-137 5 mg (Fasting) | Cohort 3: TAK-137 10 mg | Cohort 4: TAK-137 5 mg (Fasting) | Cohort 5: TAK-137 0.5 mg | Cohort 6: TAK-137 20 mg | Cohort 4: TAK-137 5 mg (Fed)
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 6
liters | 48.57 (15.521) | 62.26 (23.596) | 81.23 (47.499) | 134.49 (150.393) | 62.85 (14.652) | 110.48 (86.222) | 52.97 (17.267)

11. Secondary Outcome: Total Amount of Drug (TAK-137) Excreted in Urine From Time 0 to Time t (Ae[0-t])
Description: Total amount of drug excreted in urine from time 0 to time t, calculated as Sum (Cu*Vu), where Cu is the concentration of drug excreted in urine and Vu is the volume of urine excreted.
Time Frame: Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Cohort 1: TAK-137 2 mg | Cohort 2: TAK-137 5 mg (Fasting) | Cohort 3: TAK-137 10 mg | Cohort 4: TAK-137 5 mg (Fasting) | Cohort 5: TAK-137 0.5 mg | Cohort 6: TAK-137 20 mg | Cohort 4: TAK-137 5 mg (Fed)
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 6
mg | 0.0039 (0.00161) | 0.0164 (0.01492) | 0.0470 (0.04281) | 0.0192 (0.01465) | 0.0002 (0.00034) | 0.0585 (0.04417) | 0.0217 (0.01335)

12. Secondary Outcome: Fraction of TAK-137 Excreted in Urine (Fe)
Description: Fraction of drug excreted in urine, calculated as Fe=(Ae[0-t]/dose)×100.
Time Frame: Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent excreted
Arm/Group | Cohort 1: TAK-137 2 mg | Cohort 2: TAK-137 5 mg (Fasting) | Cohort 3: TAK-137 10 mg | Cohort 4: TAK-137 5 mg (Fasting) | Cohort 5: TAK-137 0.5 mg | Cohort 6: TAK-137 20 mg | Cohort 4: TAK-137 5 mg (Fed)
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 6
percent excreted | 0.19 (0.080) | 0.33 (0.298) | 0.47 (0.428) | 0.38 (0.293) | 0.04 (0.068) | 0.29 (0.221) | 0.43 (0.267)

13. Secondary Outcome: Renal Clearance (CLr) for TAK-137
Description: CLr is a measure of apparent clearance of the drug from the urine, calculated as CLr=Ae(0-t)/AUC(0-96).
Time Frame: Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: liters/hour
Arm/Group | Cohort 1: TAK-137 2 mg | Cohort 2: TAK-137 5 mg (Fasting) | Cohort 3: TAK-137 10 mg | Cohort 4: TAK-137 5 mg (Fasting) | Cohort 5: TAK-137 0.5 mg | Cohort 6: TAK-137 20 mg | Cohort 4: TAK-137 5 mg (Fed)
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 6
liters/hour | 0.0093 (0.00268) | 0.0094 (0.00577) | 0.0138 (0.00477) | 0.0164 (0.00626) | 0.0031 (0.00500) | 0.0117 (0.00453) | 0.0150 (0.00804)

ADVERSE EVENTS:
Time Frame: Day 1 to 14 days after the last dose of study medication (Up to 30 days).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TAK-137 0.5 mg | TAK-137 2 mg | TAK-137 5 mg (Fasting) | TAK-137 10 mg | TAK-137 20 mg | Placebo Fasting | TAK-137 5 mg (Fed) | Placebo (Fed)
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/11 | 0/6 | 0/6 | 0/12 | 0/6 | 0/2
Other Adverse Events (participants affected / at risk) | 0/6 | 1/6 | 0/11 | 1/6 | 3/6 | 4/12 | 1/6 | 0/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-137 0.5 mg (N=6) | TAK-137 2 mg (N=6) | TAK-137 5 mg (Fasting) (N=11) | TAK-137 10 mg (N=6) | TAK-137 20 mg (N=6) | Placebo Fasting (N=12) | TAK-137 5 mg (Fed) (N=6) | Placebo (Fed) (N=2)
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Orthostatic heart rate response increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.